CLINICAL TRIAL: NCT01612611
Title: A Registry Study on Safety Surveillance of Shenmai (a Chinese Medicine Injection) Used in China
Brief Title: Safety Study of Shenmai(a Chinese Medicine Injection) Used in Hospitals in China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy Director, China Academy of Chinese Medical Sciences
Other Study IDs: RSCMI-Ⅵ
Record Dates: First submitted 2012-06-03; First posted 2012-06-06 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Shock; Coronary Heart Disease
MeSH Terms: conditions — Shock; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- a cohort using Shenmai injection

SUMMARY:
The purpose of this study is to make a cohort event monitoring to see whether and how Shenmai injection in hospital results in adverse events or adverse drug reactions.

DETAILED DESCRIPTION:
Safety surveillance on Chinese Medicine injection is an important problem that needs to be sorted out ,because in mainland China hospitals ,Chinese Medicine Injection are used widely. Population for taking medicine characteristics,the incidence rate of ADR and other uncertain factors influence can not be found now.

A registry study for shenmai injection safety surveillance with 30000 patients will be conducted from Jan.2012 to Dec.2015.

Eligibility criteria Patients who will use shenmai injection in selected hospitals.

ELIGIBILITY:
Inclusion Criteria:

* all inpatients use Shenmai injection in 30 selected hospitals during their hospital stay

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all inpatients used Shenmai injection in 30 selected hospitals in mainland China
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2012-01; Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yan M Xie, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences
Locations (1):
- Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China